CLINICAL TRIAL: NCT02862431
Title: A Double-Blind, Randomized, Placebo-Controlled, Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-64565111 in Men and Women With Type 2 Diabetes Mellitus
Brief Title: Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-64565111 in Type 2 Diabetes Mellitus (T2DM)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: manufacturing-related issues
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108166; 64565111EDI1001 (Other: Janssen Research & Development, LLC); 2016-001084-37 (EudraCT Number)
Record Dates: First submitted 2016-06-24; First posted 2016-08-11 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (JNJ-64565111 2.5 nmol/kg or Placebo) (Experimental): Participants in ratio of 3:1 will receive 2.5 Nanomole Per Kilogram (nmol/kg) JNJ-64565111 or placebo.
  Interventions: Drug: JNJ-64565111; Drug: Placebo
- Cohort 2 (JNJ-64565111 3 nmol/kg or Placebo) (Experimental): Participants in ratio of 3:1 will receive 3.0 nmol/kg JNJ-64565111 or placebo. Dose may be escalated based on review by Sponsor and Principal Investigator of blinded safety, tolerability, pharmacokinetic, and (all available) pharmacodynamic data collected up to Day 29 but dose will not exceed 3.5 nmol/kg.
  Interventions: Drug: JNJ-64565111; Drug: Placebo
- Cohort 3 (JNJ-64565111 3.5 nmol/kg or Placebo) (Experimental): Participants in ratio of 3:1 will receive 3.5 nmol/kg JNJ-64565111 or placebo. Dose may be escalated based on review by Sponsor and Principal Investigator of blinded safety, tolerability, pharmacokinetic, and (all available) pharmacodynamic data collected up to Day 29 but dose will not exceed 3.5 nmol/kg.
  Interventions: Drug: JNJ-64565111; Drug: Placebo
- Cohort 4 (JNJ-64565111 Repeat or Lower Dose or Placebo) (Experimental): Participants in ratio of 3:1 will receive a dose of JNJ-64565111 or placebo that would be a repeat or lower dose level previously assessed as well-tolerated.
  Interventions: Drug: JNJ-64565111; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-64565111 — Participants will receive JNJ-64565111 subcutaneously in the abdomen on Days 1, 8, 15 and 22.
Drug: Placebo — Participants will receive Placebo subcutaneously in the abdomen on Days 1, 8, 15 and 22.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of JNJ-64565111 in adult Men and Women (of non-child bearing potential) with Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes Mellitus (T2DM) at least 3 months prior to Screening
* On a stable treatment regimen at least 3 months prior to Screening of (1) diet and exercise, or (2) metformin monotherapy (at a dose of at least 1,000 milligram (mg) per day)
* Blood pressure between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and between 60 and 100 mmHg diastolic, inclusive at Screening (sitting) and Day -2 (supine). If blood pressure is out of range, up to 2 repeated assessments are permitted
* HbA1c greater than or equal to 6.5% and less than 8.5% at Screening
* Females of non-childbearing potential

Exclusion Criteria:

* History of, or currently active, significant illness or medical disorders, including cardiovascular disease (including cardiac arrhythmias, myocardial infarction, stroke, peripheral vascular disease), hematological disease (example, von Willebrand's disease or other bleeding disorders), respiratory disease, hepatic or gastrointestinal disease, neurological or psychiatric disease, ophthalmologic disorders, neoplastic disease, skin disorder, renal disorder, or any other illness that the Principal Investigator (PI) considers should exclude the participant or that could interfere with the interpretation of the study results
* Previous surgical treatment for obesity (example, gastric bypass, gastric banding)
* History of diabetic neuropathy with signs of gastroparesis and/or known proliferative retinopathy or maculopathy
* History or current diagnosis of acute or chronic pancreatitis
* History of an invasive cardiovascular surgical procedure including, but not limited to, coronary artery bypass graft (CABG), or percutaneous coronary intervention (PCI)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2016-11-29 (Actual); Study Completion 2016-12-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Up to Day 72

SECONDARY OUTCOMES:
Number of Participants With Incidence of Anti-JNJ-64565111 Antibodies as Measure of Immunogenicity | Up to Day 72
Change From Baseline in Body Weight | Baseline, up to Day 72
Maximum Observed Plasma Concentration (Cmax) | Up to Day 72
  Maximum observed plasma concentration (Cmax) will be assessed after first dose and last dose.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Up to Day 72
  Tmax defined as actual sampling time to reach maximum observed analyte concentration will be assessed after first dose and last dose.
Area Under Concentration from time zero to the last quantifiable concentration AUC(0-last) | Up to Day 72
  AUC from time zero to the last quantifiable concentration will be assessed after first dose and after last dose.
Area Under Curve over the dosing interval AUC(0-tau) | Up to Day 72
  The AUC [0-tau] is the measure of the plasma drug concentration from time zero to end of dosing interval. It is used to characterize drug absorption. AUC [0-tau] will be assessed after first dose and last dose.
Elimination Half-Life (t1/2) | Up to Day 72
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. t1/2 will be assessed after first dose and last dose.
Apparent Clearance (CL/F) | Up to Day 72
  The Oral Clearance (CL/F) is the clearance based on oral bioavailability. CL/F will be assessed after first dose and last dose.
Apparent Volume of Distribution (V/F) | Up to Day 72
  Apparent volume of distribution will be assessed after first dose and last dose.
Terminal Rate Constant (K) | Up to Day 72
  Terminal rate constant will be assessed after first dose and last dose.
Average concentration over the dosing interval at steady state (Caverage,ss) | Up to Day 72
  The average concentration over the dosing interval at steady state, calculated as AUC(0-tau)/tau and will be assessed after last dose.
Minimum Observed Plasma Concentration (Cmin) | Up to Day 72
  The Cmin is the minimum observed plasma concentration over the dosing interval at steady state. Cmin will be assessed after last dose.
Area Under Curve from time zero extrapolated to infinity AUC(0-inf) | Up to Day 72
  AUC from time zero extrapolated to infinity will be assessed after last dose.
Accumulation Ratio | Up to Day 72
  Accumulation ratio calculated as AUC(0-tau), Day 22 / AUC(0-tau), Day 1 will be assessed after last dose.
Change From Baseline in Blood Pressure | Baseline, up to Day 72
Change From Baseline in Heart Rate | Baseline, up to Day 72
Change From Baseline for 24-hour Mean Plasma Glucose | Baseline, Day 26
  Mean plasma glucose defined as the total and/or incremental area under the concentration (AUC) time curve over 0 to 24 hours, divided by 24.
Change From Baseline in Fasting Plasma Glucose (FPG) | Baseline, up to Day 72
Change From Baseline in Hemoglobin A1c (HbA1c) | Baseline, up to Day 72
Change From Baseline on Fasting Lipids | Baseline, up to Day 72
  Total cholesterol, low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), very low-density lipoprotein cholesterol (VLDL-C), triglycerides and free fatty acids will be reported.
Change From Baseline in Insulin Secretion | Baseline, Day 26
Change From Baseline in Insulin Sensitivity | Baseline, Day 26
Change From Baseline for C-peptide | Baseline, Day 26
Change From Baseline for Glucagon | Baseline, Day 26

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Neuss, Germany